CLINICAL TRIAL: NCT05671354
Title: The Acceptability of Auto-wrapping Commode Chair in Elderly Residential Setting: A Single Group Pre-post Study
Brief Title: The Acceptability of Auto-wrapping Commode Chair in Elderly Residential Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Haven of Hope Hospital (Other); The Social Innovation and Entrepreneurship Development Fund, Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Derek Yee-Tak Cheung, Principal Investigator, Assistant Professor, The University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HKU_commode_protocol_v1
Record Dates: First submitted 2023-01-02; First posted 2023-01-04 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Technology
Keywords: Toilet hygiene; Excretions; Gerontechnology

STUDY DESIGN:
Intervention Model Description: The participants will be trained by the care staff to use the auto-wrapping commode chair. They will use the auto-wrapping commode chair for 7 days. The auto-wrapping commode chairs will seal off the excretions in a plastic bag when a button is pressed, and then prepare a new bag for next excretions. The sealed excretions will then be disposed of as usual garbage. The same staff, who are responsible for disposing of the excretions from the commodes in the previous 7 days before the trial, will dispose of the excretions from the auto-wrapping commode chairs during the trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The auto-wrapping commode chair (Experimental): The experimental group will use the auto-wrapping commode chair for 7 days.
  Interventions: Device: the auto-wrapping commode chair

INTERVENTIONS:
Device: the auto-wrapping commode chair — The auto-wrapping commode chairs will seal off the excretions in a plastic bag when a button is pressed, and then prepare a new bag for next excretions. The sealed excretions will then be disposed of as usual garbage. The same staff, who are responsible for disposing of the excretions from the commodes in the pre-test, will dispose of the excretions from the auto-wrapping commode chairs during the trial.

SUMMARY:
The study has 4 research questions regarding the use of auto-wrapping commode chairs in elderly residential setting:

Primary study questions:

1. Can the frequency of the spills of excretions during disposing of excretions be reduced when auto-wrapping commode chairs are used as compared to conventional commode chairs?

   Auxiliary study questions:
2. Can the staff time spent on disposing of excretions from commode chairs be reduced when auto-wrapping commode chairs are used as compared to conventional commode chairs?
3. What is the satisfaction of the residents and staff on using the auto-wrapping commode chairs?
4. What are the perceived benefits and feasibility in allowing the residents to use the auto-wrapping commode chairs?

DETAILED DESCRIPTION:
Study design

The trial is a single group pre-post study at Haven of Hope Woo Ping Care & Attention Home. Ten residents, who use conventional commode chair for at least 7 days before the trial, will use the auto-wrapping commode chair for 7 days. Qualitative interviews will be conducted with the participants and related staff after the participants finish using the auto-wrapping commode chair.

This protocol complies with the International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use - Guideline for Good Clinical Practice (ICH-GCP) and Declaration of Helsinki.

Subjects

Residents of 3 different floors in Haven of Hope Woo Ping Care & Attention Home and their related care staff will be recruited.

Inclusion criteria of the residents:

* Use conventional commode chair at the bedside for at least 7 days before the trial, or
* Use diapers and is suitable to use auto-wrapping commode chairs, as assessed by a nurse

Inclusion criteria of the staff:

• Are responsible for assisting toileting of the participants, including disposing of excretions

Exclusion criteria of the residents and staff:

• None

Procedures

1. Training of care staff Care staff will be trained on how to dispose of the excretions from the auto-wrapping commode chairs and facilitate the participants to use the auto-wrapping commode chairs. The training will last for around half an hour. A protocol including related operation will be provided for care staff.
2. Participants' recruitment and consent The care staff and nurses will check the eligibility of the residents and invite eligible residents to join the trial. Residents scoring above the cutoff for dementia in Montreal Cognitive Assessment (MoCA) (see Appendix 1) and not receiving a medical diagnosis of dementia or other mentally incapacitating disease will be classified as competent in giving consent and will be invited to give consent. For residents scoring below the cutoff in MoCA or receiving a diagnosis of mentally incapacitating disease, the criteria stated in the Alzheimer Europe Report (2011) will be followed to ensure that they are provided chances to give consent. In particular, four criteria will be evaluated, including 1) the person must have sufficient capacity to understand the information, 2) the person is able to retain, use and weight up such information for making a decision, 3) the person will understand the benefit, risk, and convenience, 4) the person must have the ability to communicate the decision. The University of Hong Kong (HKU) research staff and the care staff will first commit them in a causal chat to assess their ability to communicate and understand the dialogues.

   If residents are competent in giving consent, both residents and their family members will be approached for consent. In cases residents are not competent in giving consents, only their family members will be approached for consent. They will then be referred to join a 1-to-1 study introduction session. In this session, HKU research staff and service unit staff will introduce the study to the participant, and invite them to sign a consent form. As a voluntary participation, the participants have the right to withdraw from the study and intervention any time without consequences.

   Staff's consent will be sought when they are interviewed about the perceived benefits and feasibility in allowing the residents to use the auto-wrapping commode chairs.
3. Pre-test Before the use of the auto-wrapping commode chairs, there will be a 7-day pre-test. During pre-test, at regular times of the day, the standard procedure of disposing of the excretions from conventional commode chairs will be followed. This procedure includes transporting the bedpans of the commode chairs to the toilets, disposing of the excretions into the toilets, and finally transporting these bedpans to cleaning machines.

   In this period, the care staff will record daily the frequency of the spills of excretions during disposing of excretions from participants' conventional commode chairs (including transporting and disposing of the excretions to the toilets). The time spent on disposing of excretions from the conventional commode chairs will be calculated by multiplying daily frequency of disposing of excretions and average duration of disposing of excretions. Daily frequency of disposing of excretions will be retrieved from care routine schedule. Average duration of disposing of excretions will be estimated by three observations of the process by a HKU research assistant.

   In the same pre-test period, the staff will rate daily two items on the satisfaction of the participants in using, and the staff in allowing the participants to use conventional commode chairs on a 5- point Likert scale (1 = very unsatisfied; 5 = very satisfied).
4. Trial period The participants will be trained by the care staff to use the auto-wrapping commode chair. They will use the auto-wrapping commode chair for 7 days. The auto-wrapping commode chairs will seal off the excretions in a plastic bag when a button is pressed, and then prepare a new bag for next excretions. The sealed excretions will then be disposed of as usual garbage. The same staff, who are responsible for disposing of the excretions from the commodes in the previous 7 days before the trial, will dispose of the excretions from the auto-wrapping commode chairs during the trial.

During the trial, the staff will record daily the frequencies of spills of excretions during disposing of excretions as well as the satisfaction of the participants and the staff to use auto-wrapping commode chairs. The time spent on disposing of excretions from the auto-wrapping commode chairs will be calculating by multiplying daily frequency of disposing of excretions and average duration of disposing of excretions. Daily frequency of disposing of excretions will be retrieved from care routine schedule. Average duration of disposing of excretions will be estimated by three observations of the process by a HKU research assistant.

Qualitative interviews will be conducted with all participants when they finish using the auto-wrapping commode chairs. 2-3 related staff of each site will be interviewed after all participants complete or terminate the trial. Interview contents include the perceived benefits and feasibility in allowing the residents to use the auto-wrapping commode chairs as compared to conventional commode chairs.

Blinding

No blinding will be done for this single group study.

Sample size determination

The sample size is estimated by the expected number of eligible residents of the sites. A maximum of 10 participants will be recruited from each site.

Data analysis

1. Main analysis Wilcoxon signed-rank test will be used to examine the difference in the frequency of the spills of excretions during disposing of excretions between using auto-wrapping commode chairs and conventional commode chairs, and the difference in the staff time spent on disposing of excretions from auto-wrapping commode chairs and conventional commode chairs.

   Descriptive statistics will be used to explore the satisfaction on the auto-wrapping commode chairs.
2. Qualitative interview The qualitative interview content will be transcribed verbatim in Chinese for further analysis. The qualitative interview transcripts will then be analyzed using framework analysis to construct a coherent and logical structure from the classification of many opinions and perceptions of the new health monitoring device. The results will then be discussed and consolidated in the panel meetings with the co-authors.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria of the residents:

* Use conventional commode chair at the bedside for at least 7 days before the trial, or
* Use diapers and is suitable to use auto-wrapping commode chairs, as assessed by a nurse

Inclusion criteria of the staff:

• Are responsible for assisting toileting of the participants, including disposing of excretions

Exclusion Criteria:

Exclusion criteria of the residents and staff:

• None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2023-03-05 (Actual); Primary Completion 2023-05-03 (Actual); Study Completion 2023-05-03 (Actual)

PRIMARY OUTCOMES:
The frequency of the spills of excretions during disposing of excretions from the conventional and auto-wrapping commode chairs. | 7 days before the 7-day trial period to the end of the 7-day trial period
  The frequency of the spills of excretions during disposing of excretions from the conventional commode chairs will be recorded by the care staff at the end of night shifts during 7 days before the 7-day trial period. The frequency of the spills of excretions during disposing of excretions from the auto-wrapping commode chairs will be recorded by the care staff at the end of night shifts during the 7-day trial period.

SECONDARY OUTCOMES:
The staff time spent on disposing of excretions from conventional and auto-wrapping commode chairs | 7 days before the 7-day trial period to the end of the 7-day trial period
  The staff time spent on disposing of excretions from conventional and auto-wrapping commode chairs will be recorded by a HKU research assistant during two demonstration sessions. In one demonstration session before the 7-day trial period, the care staff will demonstrate the procedures of disposing of excretions from conventional commode chairs for 3 times, and the time will be recorded by a HKU research assistant. In one demonstration session during the 7-day trial period, the care staff will demonstrate the procedures of disposing of excretions from auto-wrapping commode chairs for 3 times, and the time will be recorded by a HKU research assistant.
The satisfaction of the residents and staff on using conventional and auto-wrapping commode chairs | From the start to the end of the 7-day trial period
  The satisfaction of the residents and staff on using conventional commode chairs will be recorded by the care staff at the end of night shifts during 7 days before the 7-day trial period. The satisfaction of the residents and staff on using auto-wrapping commode chairs will be recorded by the care staff at the end of night shifts during the 7-day trial period.
Qualitative measure: The perceived benefits and feasibility in allowing the residents to use the auto-wrapping commode chairs as compared to conventional commode chairs and toilets. | At the end of the 7-day trial period
  Qualitative interviews will be conducted with all participants when they finish using the auto-wrapping commode chairs. 2-3 related staff of each site will be interviewed after all participants complete or terminate the trial. Interview contents include the perceived benefits and feasibility in allowing the residents to use the auto-wrapping commode chairs as compared to conventional commode chairs.

CONTACTS AND LOCATIONS:
Overall Officials: Yee Tak Cheung, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- Haven of Hope Woo Ping Care & Attention Home, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Research data and documentation will be available upon request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available for 10 years.